CLINICAL TRIAL: NCT04261751
Title: Validation of the Moral Injury Symptom Scale Clinician Version Short Form and Moral Injury Outcome Scale in Nurses
Brief Title: Moral Injury Symptom Scale/Moral Injury Outcome Scale
Acronym: MISS MIOS
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1497904
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Moral Injury; Anxiety; Depression; Burn-Out
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses: Nurses will be taking the Clinician Questionnaire electronically.
  Interventions: Other: Clinician Questionnaire

INTERVENTIONS:
Other: Clinician Questionnaire — Nurses will take the Clinician Questionnaire electronically

SUMMARY:
The purpose of this research is to validate the moral injury symptom scale clinician version short form and the Moral Injury Outcome Scale in nurses. Participants will be recruited in accordance with AdventHealth Policy # 400.120: Selection and Enrollment of AdventHealth Employees, Physicians, and Volunteers for research Studies. Employee participants will be assured participation in this study will not affect performance evaluation or employment-related decisions by peers or supervisors. No employees will be recruited by a direct supervisor. Recruitment of potential employees as participants will occur without coercion by the Principal Investigator (PI), by bulletin board advertisements, or through a third party unassociated in a power/supervisory relationship with the employee (i.e., researchers from Center for Whole-Person Research).

ELIGIBILITY:
Inclusion Criteria:

1. Currently working as a registered nurse (Licensed Practical Nurse, Registered Nurse, Assistant Nurse Manager, Nurse Manager, Nurse Educator) at identified hospital within the state of Florida
2. Access to computer or mobile device to complete the survey
3. Ability to read and understand English

Exclusion Criteria:

1. Any employee at identified hospitals who is not a licensed nurse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Licensed nurses at identified hospital within the state of Florida
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Moral Injury | 1 Day
  measured by the Moral Injury Outcome Scale & functional outcomes (23 items), and the Moral Injury Symptom Scale - Clinician Version - Short Form (MISS-CV-SF) 11 items. The scale is 10 - 100 with the higher number being worse.

SECONDARY OUTCOMES:
Spiritual Wholeness | 1 Day
  measured by Spiritual Wholeness Screening 4 items (yes/no)
Social involvement/Social Support | 1 Day
  measured by 1 social support/social involvement item
Depression | 1 day
  measured by the PhQ-9 Depression scale (9 items)
Burnout | 1 Day
  measured by Stanford Professional Fulfillment Index (16 items), and the MBI (22 items)
Anxiety | 1 Day
  measured by GAD-7 (7 items)
Spiritual Well Being | 1 Day
  measured by FACIT-SP (12 items)
Moral injury | 1 Day
  measured by the Moral Injury Events Scale (9 items) and the Expressions of Moral Injury Scale (17 items)
PTSD | 1 Day
  measured by PCL-5 (20 items)
Post-traumatic growth | 1 Day
  measured by Post-Traumatic Growth Inventory (21 items0
Nurse Job Satisfaction | 1 Day
  measured by the Nurse Job Satisfaction Scale (10 items)
Satisfaction with care/time demands | 1 Day
  measured by 1 item
Prevalence of aggression | 1 Day
  measured by Perception of Prevalence of Aggression Scale (adapted) 11 items
Discrimination | 1 Day
  measured by Everyday Discrimination Scale (10 items)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Tao, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No